CLINICAL TRIAL: NCT06973148
Title: Evaluation of Oxidative Stress and Methylated Arginine Levels in Individuals With Periodontitis
Status: Completed | Type: Observational
Sponsor: Ankara Medipol University (Other)
Collaborators: Ankara University (Other); Medipol University (Other)
Responsible Party: Principal Investigator, Zeliha Guney, Assoc. Prof., Ankara Medipol University
Other Study IDs: 04/11; 17.02.2021, 04/11 (Other: the Human Research Ethics Committee of Ankara University)
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Oxidative Stress
Keywords: periodontitis; oxidative stress; antioxidante; methylated arginines
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- periodontitis group: Stage III Grade B periodontitis
- Healthy group: periodontally healthy

SUMMARY:
You are being invited to participate in a scientific research study. Before you decide to take part, it is essential that you understand why the study is being conducted and what your participation will involve. Please take the time to read the following information carefully. Feel free to ask if anything is unclear or need more details.

This study aims to evaluate saliva composition, specifically focusing on amino acid and protein building blocks, oxidative stress, and the Nitric Oxide metabolism system, including levels of ADMA (Asymmetric Dimethylarginine) and SDMA (Symmetric Dimethylarginine). By examining these parameters, we aim to contribute to a better understanding of the biological mechanisms involved in gum health and systemic responses.

You have been selected to participate in this study based on your periodontal (gum) health status. A total of 40 individuals, 20 diagnosed with periodontitis and 20 diagnosed as periodontally healthy, who meet the study criteria, will be included.

If you choose to participate, you will receive non-surgical periodontal treatment as part of your routine care. Before the treatment, biological samples, including saliva and serum, will be collected. These samples will be used solely for scientific analysis and will not affect the outcome of your dental treatment. Although the total duration of the study is 2 years, your involvement will conclude at the beginning of periodontal therapy.

There are no anticipated risks associated with participation beyond those commonly encountered during dental examinations and treatments. You will not benefit directly; however, your contribution will help advance scientific knowledge about the factors influencing oral and systemic health.

All information collected from you during the study will remain confidential. Your identity will be protected, and personal data will not be disclosed in any reports or publications resulting from this study.

Participation in this study is entirely voluntary. You are free to decline or withdraw at any time, without needing to give a reason. Your decision will not affect the quality of care you receive.

All tests, examinations, and procedures performed as part of this study will be provided at no cost to you. Participation will not result in any financial cost or compensation.

DETAILED DESCRIPTION:
This scientific research study is designed to investigate the biological components of saliva, with particular attention to specific biomarkers related to gum health and broader systemic functions. The study focuses on evaluating amino acids and protein building blocks in saliva, markers of oxidative stress, and elements of the Nitric Oxide metabolism system. Special emphasis is placed on measuring the levels of Asymmetric Dimethylarginine (ADMA) and Symmetric Dimethylarginine (SDMA), which are known to play roles in vascular and inflammatory processes.

The primary objective is to enhance understanding of the biological mechanisms that underpin periodontal (gum) health and disease, as well as to explore potential systemic interactions. By comparing biological parameters between individuals with periodontitis and those who are periodontally healthy, the study seeks to identify patterns and correlations that may inform both preventive and therapeutic strategies in dental care and possibly broader health contexts.

The study will enroll a total of 40 participants, divided equally between two groups:

* 20 individuals diagnosed with periodontitis.
* 20 individuals diagnosed as periodontally healthy.
* Participants are selected based on their periodontal health status and must meet specific inclusion criteria set by the research team.

Participation Process:

Participants will undergo standard, non-surgical periodontal treatment as part of their regular dental care.

Prior to the commencement of this treatment, biological samples, including saliva and blood serum, will be collected.

These samples are used strictly for scientific purposes and will not interfere with the participants' clinical care or treatment outcomes.

The study itself spans a period of 2 years, but the participants' active involvement is limited to the time up to the start of their periodontal therapy.

Risks and Benefits:

The study is considered low-risk. The procedures involved do not present risks beyond those typically associated with standard dental examinations and treatments.

Participants will not receive direct personal benefit from the study. However, their involvement will significantly contribute to advancing scientific knowledge in the fields of periodontology and systemic health.

Confidentiality and Data Protection:

All information gathered during the study will be handled with strict confidentiality.

Personal identifiers will be removed or coded to ensure anonymity in any reports or publications.

Data protection measures will comply with ethical standards and legal requirements.

Voluntary Participation:

Participation is entirely voluntary. Participants have the right to refuse or withdraw from the study at any point, without providing a reason.

Withdrawal will not affect the standard or quality of care provided.

Financial Considerations:

There is no cost to participants for any procedures or tests carried out as part of the study.

No financial compensation will be provided for participation. In summary, this study is a scientific endeavor aimed at deepening understanding of the biological links between periodontal health and broader systemic markers, with no expected harm or direct benefit to the participants, and with all necessary ethical safeguards in place.

ELIGIBILITY:
Inclusion Criteria:

* Having at least 16 natural teeth
* Aged between 18 and 64 years
* Systemically healthy (no known systemic diseases)

Exclusion Criteria:

* Having diabetes, cancer, cardiovascular diseases, and/or any autoimmune diseases such as rheumatoid arthritis
* Pregnant and lactating mothers 3-Tobacco users
* Patients using antibiotics, anti-inflammatory medications, immunosuppressive drugs, and contraceptives within three months
* Patients who had periodontal treatment during the last six months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of individuals recruited from the Department of Periodontology, Ankara University Faculty of Dentistry, between June 2021 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Power analysis | Baseline
  Sample size analysis was performed a priori using G*Power software before the initiation of the study. The analysis applied a large effect size (Cohen's d = 0.8) for independent two-group comparisons, with a significance level (α) of 0.05 and a statistical power of 80%, resulting in a calculated total sample size of 40 participants.
Plaque Index (PI) | Baseline
  Separate intergroup comparisons will be conducted for each clinical outcome measure to allow precise and independent reporting. Thea plaque index (PI), assessed using the Silness and Löe plaque index, which evaluates the thickness of plaque along the gingival margin on a scale from 0 (no plaque) to 3 (abundant plaque). All cl
Probing depth (PD) | Baseline
  The probing depth (PD), measured in millimeters at six sites per tooth (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual) using a standardized manual periodontal probe (e.g., UNC-15 probe) with markings at 1 mm increments to ensure accuracy.
Bleeding on probing (BOP) | Baseline
  The bleeding on probing (BOP), recorded as the presence or absence of bleeding within 15 seconds of probing at each site and reported as the percentage of positive sites per participant.
Clinical attachment loss (CAL) | Baseline
  Separate intergroup comparisons will be conducted for each clinical outcome measure to allow precise and independent reporting. The clinical attachment loss (CAL), also measured in millimeters at the same six sites per tooth, calculated as the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket.
Determination of salivary and serum oxidative stress index | Baseline
  Total antioxidant status (TAS) and total oxidant status (TOS) were measured at Baseline in saliva and serum samples using Erel's validated method. TAS was based on the reduction of the ABTS⁺ (2,2'-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid)) radical by antioxidants, causing a decrease in color intensity read at 600 nm with a Varioskan Multimode Reader. Calibration used ascorbic acid; results were expressed in mmol ascorbic acid equivalents/L. Higher TAS indicates stronger antioxidant capacity. TOS involved oxidation of Fe²⁺ to Fe³⁺, forming a colored complex with xylenol orange, read at 530 nm; results were in μmol H₂O₂ equivalents/L. Higher TOS reflects elevated oxidant levels. The oxidative stress index (OSI) was calculated as (TOS/TAS) × 10, a unitless index where higher values indicate greater oxidative stress. All assays were performed in duplicate for reliability.
Determination of Salivary and Serum Methylated Arginine Metabolites | Baseline
  Salivary and serum levels of arginine, asymmetric dimethylarginine (ADMA), and symmetric dimethylarginine (SDMA) were measured at the baseline time point. Quantification was performed using liquid chromatography-tandem mass spectrometry (LC-MS/MS) with an electrospray ionization (ESI) source (Thermo Scientific Accessmax). Samples underwent protein precipitation and derivatization before injection. Chromatographic separation was achieved on a reversed-phase column under optimized gradient conditions, and mass detection was performed in multiple reaction monitoring (MRM) mode for high specificity. Calibration curves with known standards ensured quantitative accuracy, and results were expressed in micromoles per liter (µmol/L). All measurements were performed in duplicate for reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Guney, Principal Investigator — Ankara Medipol University; Sivge Kurgan, Prof., Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Balkan B, Guney Z, Balkan E, Balkan EP, Kurgan S, Balci N, Serdar MA, Gunhan M. Interaction between methylated arginine metabolites and oxidative stress in periodontitis: a cross-sectional study. BMC Oral Health. 2025 Nov 14;25(1):1781. doi: 10.1186/s12903-025-06972-6. PMID 41239382